CLINICAL TRIAL: NCT04256980
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib in Subjects With Advanced/Metastatic or Surgically Unresectable Cholangiocarcinoma Including FGFR2 Rearrangement Who Failed at Least One Previous Therapy
Brief Title: Pemigatinib in Treating Patients With Advanced/Metastatic or Surgically Unresectable Cholangiocarcinoma Including FGFR2 Rearrangement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI375A201
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cholangiocarcinoma
Keywords: CCA; FGFR2; Pemigatinib
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pemigatinib in patients with advanced/metastatic or surgically (Experimental): Patients with advanced/metastatic or surgically unresectable cholangiocarcinoma
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib will be self-administered at 9mg Or 13.5mg as a QD oral treatment on a 2-week-on therapy and 1-week-off therapy schedule

SUMMARY:
This is a phase 2 study to investigate the efficacy and safety of Pemigatinib in treating patients with advanced/metastatic or surgically unresectable cholangiocarcinoma with FGFR2 rearrangement who have failed at least 1 previous therapy

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 or older.
2. Histologically or cytologically confirmed cholangiocarcinoma which was considered to be advanced/metastatic or surgically unresectable by the investigator through image examination.
3. Radiographically measurable disease per RECIST v 1.1
4. Documentation of FGFR2 rearrangement.
5. Documented disease progression after at least 1 line of prior systemic therapy.
6. ECOG performance status of 0~1.
7. Life expectancy ≥12 weeks.

Exclusion Criteria:

1. Prior receipt of a selective FGFR inhibitor.
2. History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of softy tissues ( exception: skin, kidney, tendons or vessels due to injury, disease, and aging, in the absence of systemic mineral imbalance).
3. Currently evidence of clinically significant corneal or retinal disorder confirmed by ophthalmologic examination.
4. Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives, whichever is shorter, before the first dose of study drug. Topical ketoconazole will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate per RECIST 1.1 | Every 6 weeks for the first 2 cycles and every 9 weeks thereafter through end of treatment, up to 24 months

SECONDARY OUTCOMES:
PFS（PFS= first dose to progressive disease or death） | Time from first treatment to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
DOR（DOR= time from the date of CR or PR until PD） | Every 6 weeks for the first 2 cycles and every 9 weeks thereafter through end of treatment, up to 24 months
DCR（DCR=CR + PR + stable disease） | Every 6 weeks for the first 2 cycles and every 9 weeks thereafter through end of treatment, up to 24 months
OS（OS= first dose to death of any cause） | Time from first treatment to the date of death from any cause, up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi GM, Huang XY, Wen TF, Song TQ, Kuang M, Mou HB, Bao LQ, Zhao HT, Zhao H, Feng XL, Zhang BX, Peng T, Zhang YB, Li XC, Yu HS, Cao Y, Liu LX, Zhang T, Wang WL, Ran JH, Liu YB, Gong W, Chen MX, Cao L, Luo Y, Wang Y, Zhou H, Yang GH, Fan J, Zhou J. Pemigatinib in previously treated Chinese patients with locally advanced or metastatic cholangiocarcinoma carrying FGFR2 fusions or rearrangements: A phase II study. Cancer Med. 2023 Feb;12(4):4137-4146. doi: 10.1002/cam4.5273. Epub 2022 Sep 20. PMID 36127767